CLINICAL TRIAL: NCT05729230
Title: Evaluation of the Patient-physician Relationship During the Initial Consultation Prior to the Introduction of a New Systemic Treatment for Advanced Hepatocellular Carcinoma: Information Needs, Prognostic Awareness, Treatment Expectations Regarding Efficacy and Side Effects
Brief Title: PAtient-PHYsician Relationship Assessment
Acronym: PAPHYRA
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); ASZ Aalst (Other); Grand Hôpital de Charleroi (Other); AZ Sint-Jan AV (Other); CHC Montlegia (Other)
Responsible Party: Sponsor
Other Study IDs: P2020/448
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: systemic treatment
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Questionnaire — Physician/data nurse and the patients will complete a questionnaire. The physician or data nurse must complete a descriptive form including the patient's age and gender as well as some information about the tumour and the underlying liver disease.
  Based on the 4 open questions, patient will be classified into 2 groups after assessment of his answers by a group of digestive oncologists and psychologists. Group A includes patients with an accurate perception of the disease whereas group B will gather patients with unrealistic expectations. Psychosocial aspect, quality of the physician's communication, comprehension of the disease and treatment expectations are assessed by multiple-choice questions (Liker scale evaluation). Depression and anxiety were evaluated by the Hospital Anxiety and Depression Scale (HADS) that has been validated as a good scale with a high sensitivity and specificity for depression and anxiety for cancer patients.

SUMMARY:
I) Introduction Patients with cancer face difficult choices that require balancing competing priorities such as survival, functional capacity and symptom relief. Most patients with advanced cancer (>80%) expect frank yet sensitive discussions with their physicians about prognosis and treatment choices in order to be involved in the decision-making process. Nevertheless, this kind of discussion is frequently lacking, and consequently, patients often have a biased view of their own prognosis such as an underestimation of disease severity, or unrealistic expectations for cure.

Patients with advanced hepatocellular carcinoma (HCC) may be treated with systemic therapies which may prolong survival but are not curative. Patients with advanced HCC often report expectations for survival and treatment-related side effects that differ from their treating physician. Accordingly, communication on prognostic and treatment choices is essential to obtain an accurate understanding of the disease that allows patients to make informed decisions. To the best of our knowledge, a thorough evaluation of the physician-patient communication quality has never been performed in advanced HCC patients.

The aim of our study is to assess the perception of the expected prognosis and treatment side effects by the patient and his physician during the first consultation before the initiation of a new systemic therapy.

II) Type of study:

Prospective, observational, non-interventional multicentric study

III) Outcomes III.1) Primary Outcome Evaluate the concordance between the patient's perception of his prognosis and treatment side effects with the one of his treating physician.

III.2) Secondary Outcomes

* Compare the patient's expectations for the aforementioned items to those of his physician and the degree of concordance between them.
* Evaluation of patient satisfaction with the information received during the consultation
* Assessment of patient-reported symptoms of anxiety and depression
* Evaluate the association between individual prognosis expectation (i.e., patient and physician) and data from the available literature.

IV) Recruitment All consecutive patients with a new systemic treatment prescribed for HCC in participating centres will be included for a period of 1 year.

DETAILED DESCRIPTION:
Patients with cancer face difficult choices that require balancing competing priorities such as survival, functional capacity and symptom relief. Most patients with advanced cancer (>80%) expect frank yet sensitive discussions with their physicians about prognosis and treatment choices in order to be involved in the decision-making process. Nevertheless, this kind of discussion is frequently lacking, and consequently, patients often have a biased view of their own prognosis such as an underestimation of disease severity, or unrealistic expectations for cure.

Patients with advanced hepatocellular carcinoma (HCC) may be treated with systemic therapies which may prolong survival but are not curative. Patients with advanced HCC often report expectations for survival and treatment-related side effects that differ from their treating physician. Accordingly, communication on prognostic and treatment choices is essential to obtain an accurate understanding of the disease that allows patients to make informed decisions. To the best of our knowledge, a thorough evaluation of the physician-patient communication quality has never been performed in advanced HCC patients.

The aim of our study is to assess the perception of the expected prognosis and treatment side effects by the patient and his physician during the first consultation before the initiation of a new systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* diagnose of advanced hepatocellular carcinoma by histology or radiology using the EASL criteria
* ≥ 18 years old
* willing to participate in the study, being capable of consenting and sign the informed consent
* not candidate for curative treatment or locoregional therapy
* any line systemic therapy that has been validated by the local hepatic tumor board.

Exclusion Criteria:

* Locoregional treatment combined with systemic treatment
* Pregnancy in progress
* Candidate for surgery or locoregional therapy
* Patient with state medical aid (AME)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with advanced hepatocellular carcinoma eligible for systemic treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Perception of prognosis and treatment side effects | 12 months
  Evaluate the concordance between the patient's perception of his prognosis and treatment side effects with the one of his treating physician. Use of survey completed by the patient and the doctors to assess the primary endpoint

SECONDARY OUTCOMES:
Compare the patient's expectations for the aforementioned items to those of his physician and the degree of concordance between them. | 12 months
  Use of survey completed by the patient and the doctors to assess the primary endpoint
Assessment of patient-reported symptoms of anxiety and depression | 12 months
  Use of survey completed by the patient and the doctors to assess the primary endpoint
Evaluate the association between individual prognosis expectation (i.e., patient and physician) and data from the available literature. | 12 months
  Use of survey completed by the patient and the doctors to assess the primary endpoint
Evaluation of patient satisfaction with the information received during the consultation | 12 months
  Use of survey completed by the patient and the doctors to assess the primary endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Gontran Verset, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- University Hospital Brussels, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No